CLINICAL TRIAL: NCT04096378
Title: Improving Racial Socialization Competency for Black Caregivers Through a Culturally-Informed Familial Therapeutic Intervention
Brief Title: EMBRace With Grandparents
Acronym: EMBRace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Riana Anderson, Assistant Professor, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00160402
Record Dates: First submitted 2019-09-12; First posted 2019-09-19 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Racial Discrimination; Depression; Anxiety; Stress; Trauma, Psychological
Keywords: Racial Socialization; Family Functioning; Stress and Coping
MeSH Terms: conditions — Racism; Depression; Anxiety Disorders; Psychological Trauma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMBRace Intervention Group (Experimental): Over 13 weeks, participants will engage in a pretest (week 1) 5 weekly sessions (weeks 2-6), a posttest (week 7) and a follow-up (week 13). The intervention (Engaging, Managing, and Bonding through Race: EMBRace) seeks to reduce racial trauma for both youth and caregivers and increase family functioning via psychoeducation and therapy.
  Interventions: Behavioral: EMBRace Intervention Group
- EMBRace Waitlist Group (Other): Participants will wait for thirteen weeks without receiving EMBRace or alternative therapeutic sessions. The waitlist group will subsequently become the intervention group with the opportunity to participate in the EMBRace intervention protocol above.
  Interventions: Behavioral: EMBRace Waitlist Group

INTERVENTIONS:
Behavioral: EMBRace Intervention Group — The EMBRace intervention will consist of five weekly sessions (weeks 2 - 6) that will be facilitated by EMBRace-trained therapists. Throughout the 8-week intervention, families will be scheduled for 2-hour blocks with sessions being administered to each parent and adolescent for 90 minutes (individually for 30 minutes, 15-minute break, and 45-minutes session with parent and adolescent together). The sessions will cover research-based types of Racial Socialization, including cultural pride, preparation for bias, and attentiveness and balance towards societal racism. Parents and youth will also learn and practice five literacy skills to process and manage the stress of racial encounters including the ability to recognize racial discrimination, accurately appraise the stress of self and others, reduce one's stress, engage instead of avoid, and finally resolve toward healthy outcomes.
  Arms: EMBRace Intervention Group
Behavioral: EMBRace Waitlist Group — The waitlist group will be asked to complete a pretest and posttest while the treatment group goes through the EMBRace intervention. During this time, the waitlist group will not have any additional requirements and will not be given any form of comparative treatments. Upon the completion of the treatment from the intervention group, the waitlist group will be consented for entry into the intervention arm of the study and will follow the procedures for the intervention group above.
  Arms: EMBRace Waitlist Group

SUMMARY:
Research on racial discrimination (RD) continues to show the debilitating toll on mental and physical health for adolescents throughout their developmental trajectory, particularly for Black Americans. While adolescents may employ emotion-focused behaviors (e.g., overeating, etc.) in-the-moment to reduce discriminatory distress, such risk-laden behaviors can result in later disparities in their overall health. While this link has been repeatedly established in the literature, racially-specific protective mechanisms (e.g., racial socialization; RS) have been shown to disrupt the pathway from discrimination to health-related outcomes in adolescents. Although informative, the literature on RS has yet to advance our understanding of ways to improve upon these protective processes in Black families. Thus, the proposed study will further our understanding by aiming to improve RS competency (e.g., skills and efficacy) among African American caregivers and youth (ages 10-14) in Detroit, Michigan through the Engaging, Managing, and Bonding through Race (EMBRace) intervention.

The EMBRace intervention facilitates spaces where Black caregivers strengthen and develop skills to be attentive to their adolescent's racial trauma while also reducing their own stress via racial coping knowledge and RS strategies. Parents and adolescents start each session by engaging in separate therapeutic sessions to process experiences of their Black identity. They will then join together for a family session that focuses on enhancing messages about racial pride, bias preparation, rationales behind promoting distrust, and why not engaging in RS practices may be detrimental to youth. EMBRace sessions will take place at the University of Michigan Detroit Center and community sites, and will be video recorded to improve upon the delivery of therapeutic techniques to the families we serve.

DETAILED DESCRIPTION:
Approximately 90% of Black youth report facing or witnessing racial discrimination in their proximal (e.g., classroom) and virtual (e.g., social network) environments. The association between discrimination and negative mental health outcomes (e.g., more severe and higher rates of depression) has been repeatedly established in the literature. Moreover, discrimination impairs the way youth cope, and it is this compromised coping that is associated with negative psychological, academic, and health outcomes. Further, adolescent outcomes may lead to marked health complications and widening disparities in adulthood. Within adolescence, families can have a contributing role in the buffering or exacerbation of coping processes and behaviors to discriminatory experiences. The majority of Black families use racial socialization (RS)-or the verbal and nonverbal communication regarding racial matters-to facilitate coping with race. While RS has been shown to disrupt the trajectory from discrimination to negative psychological outcomes in some respects, it has also contributed to increased youth depressive and anxious symptoms given the wide variety of strategies observed in RS communication. Furthermore, less is known about the impact that grandparents have in the socialization process of their adolescent grandchildren, even though Black grandparents are more likely to rear their grandchildren compared to other races and given current trends. To address these gaps, the emergence of a new RS theory and accompanying clinical intervention seeks to investigate and improve upon this potentially protective cultural process by improving RS competency and enhancing coping processes. The Racial Encounter Coping Appraisal and Socialization Theory (RECAST) postulates that caregivers' explicit and consistent delivery of psychoeducation-informed, skilled, and confident RS practices can reduce caregiver stress and subsequent psychological problems experienced by Black youth via greater coping self-efficacy and coping behaviors. The Engaging, Managing, and Bonding through Race (EMBRace) intervention is the application of RECAST and seeks to improve upon competent RS practices through therapeutic and empirically supported strategies. The use of culturally-relevant theory in clinical treatment is vital to Black youth's coping with specific (i.e., racial) stressors linked to long-term health and wellness outcomes. The empirical investigation of RECAST can also clarify whether aging caregivers (e.g., grandparents) develop the same competencies as other primary caregivers for an intergenerational exploration of RS practices. Thus, the goal of this study is to test the effectiveness of a unique culturally-relevant and family-based intervention developed to enhance RS competencies in Black caregivers and reduce negative psychological outcomes for adolescent children. Building on the preliminary data that I collected during the acceptability pilot testing of the EMBRace intervention in Philadelphia, the proposed study will test the mechanism of caregiver RS competency as a moderator of discrimination, coping self-efficacy, coping, and adolescent psychological outcomes.

The specific aims of the study are to:

1. improve caregiver RS competency, including a decrease in stress;
2. improve adolescents' self-reported coping strategies through enhanced coping self-efficacy; and
3. decrease adolescents' self-reported psychological problems within the EMBRace treatment group.

By posttest and 6-week follow-up, EMBRace families are hypothesized to:

1. be rated as and rate themselves as more competent in their RS practices, including less stress;
2. report more satisfactory coping and higher coping self-efficacy scores; and
3. report less psychological problems relative to pre-test and a control group.

The success of an EMBRace pilot and subsequent clinical trials can lead to its uptake by service agencies and youth-facing organizations to address the pervasive societal problem of racial discrimination for Black youth and families. The reduction of psychological harm in Black families will have a reverberating impact in various systems (e.g., school, health, residential), which can also address the persistent gaps evident in these systems (e.g., achievement, life expectancy, resource). Furthermore, I seek to have a sustainable and long-term research agenda in the improvement of patient health given the community-oriented nature of EMBRace, which partners with families and organizations and trains clinicians for both the improvement of Black family outcomes and the treatment of race-related problems.

ELIGIBILITY:
Inclusion Criteria:

* The child must be between the ages of 10-14 years.
* At least one caregiver will be primarily designated to attend sessions.
* At least one biological parent must identify or be identified as African American.
* The participant is a resident of the Detroit Metropolitan Area.
* The participant's primary language is English

Exclusion Criteria:

* Having a relative who is currently an EMBRace staff member.
* At least one of the biological parents does not identify as African American.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-05-05 (Actual); Study Completion 2023-05-05 (Actual)

PRIMARY OUTCOMES:
Change in Racial Socialization Competency | Measured in caregivers at pretest (week 1), Posttest (week 7), and 6 week follow-up (week 13)
  Racial Socialization Competency (RaSCS) consists of 28 items that include " teach my child to initiate a conversation about race with peers" and "share my emotions about my positive racial encounters." Participants will answer the following questions based on their experiences within the last year. When they do the following with their children, participants indicate A) how much they think they can; B) how prepared they are; and C) how stressed they are.
Change in Adolescent Depression | Measured in youth at pretest (week 1), Posttest (week 7), and 6 week follow-up (week 13)
  The Kutcher Adolescent Depression Scale-6 (KADS-6) is a self-report scale specifically designed to diagnose and assess the severity of adolescent depression. The abbreviated 6-item scale will be used instead of the 16 or 11 item scale. The scales identify as 0-Hardly Ever, 1- Much of the time, 2 most of the time, and 3- All of the time.
Change in Problem Behaviors | Measured in youth at pretest (week 1), Posttest (week 7), and 6 week follow-up (week 13)
  Brief Problems Monitor (BPM), is a 19-item scale designed for parents to better assess their child's Internalizing (INT), Attention Problems (ATT), Externalizing (EXT), and Total Problems (TOT). Scales comprise items from the Child Behavior Checklist for Ages 6-18 (CBCL/6-18), Teacher's Report Form (TRF), and Youth Self-Report (YSR). Statements such as "acts too young/old for his age" are accompanied by a scale of 0 (being not true), 1 (somewhat true) and 2 (very true). The items, scales, and norms are based on decades of research and practical experience, as summarized in the BPM Manual.
Change in Perception of Stress | Measured in youth and caregivers at pretest (week 1), Posttest (week 7), and 6 week follow-up (week 13)
  The Perceived Stress Scale (PSS) is a psychological instrument for measuring the perception of stress. It is a 10-item Likert-based measure of the degree to which situations in one's life are appraised as stressful. Each of the items on the PSS-10 are rated on a 5-point Likert scale, ranging from 0 (never) to 4 (very often). Items were designed to tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The scale also includes a number of direct queries about current levels of experienced stress. The PSS was designed for use in community samples with at least a junior high school education. Moreover, the questions are of a general nature and hence are relatively free of content specific to any subpopulation group. The questions in the PSS ask about feelings and thoughts during the last month. In each case, respondents are asked how often.

SECONDARY OUTCOMES:
Change in Adolescent Coping Behaviors | Measured in youth at pretest (week 1), Posttest (week 7), and 6 week follow-up (week 13)
  Adolescent Coping Orientation for Problem Experiences (A-COPE) measures adolescent coping behaviors that results from the normal adolescent stress associated with trying to create a balance between being connected to and at the same time independent from one's family. A-COPE is a 54 item self-report questionnaire used to identify coping strategies employed by adolescents. (e.g., When you face difficulties or feel tense, how often do you talk to your mother about what bothers you?) Responses of A-COPE are measured on a 5-point Likert scale (never, hardly, sometimes, often, most of the time).
Change in Adolescent Racial Distress | Measured in youth at pretest (week 1), Posttest (week 7), and 6 week follow-up (week 13)
  The Adolescent Discrimination Distress Index measures distress associated with instances of perceived racial prejudice encountered in educational contexts. It is a 15-item scale, each question asking, "Have you experienced this?" Responses are in dichotomous format with "yes/no" answer options. If answered yes, each question will ask "If you had this experience, did it upset with?" with a Likert response scale of 1-5. 1 (not at all), 2 (slightly), 3 (moderately), 4 (considerably), 5 (extremely).

CONTACTS AND LOCATIONS:
Overall Officials: Riana E Anderson, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Detroit Center, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share participants' data with other researchers.

REFERENCES:
- [Background] Anderson RE, Stevenson HC. RECASTing racial stress and trauma: Theorizing the healing potential of racial socialization in families. Am Psychol. 2019 Jan;74(1):63-75. doi: 10.1037/amp0000392. PMID 30652900
- [Result] Anderson RE, McKenny MC, Stevenson HC. EMBRace: Developing a Racial Socialization Intervention to Reduce Racial Stress and Enhance Racial Coping among Black Parents and Adolescents. Fam Process. 2019 Mar;58(1):53-67. doi: 10.1111/famp.12412. Epub 2018 Dec 15. PMID 30552778
- [Result] Anderson RE, Jones SCT, Navarro CC, McKenny MC, Mehta TJ, Stevenson HC. Addressing the Mental Health Needs of Black American Youth and Families: A Case Study from the EMBRace Intervention. Int J Environ Res Public Health. 2018 May 2;15(5):898. doi: 10.3390/ijerph15050898. PMID 29724068
- [Result] Anderson RE, McKenny M, Mitchell A, Koku L, Stevenson HC. EMBRacing racial stress and trauma: Preliminary feasibility and coping responses of a racial socialization intervention. Journal of Black Psychology 44(1): 25-46, 2018.